CLINICAL TRIAL: NCT06384781
Title: Development, Refinement, and Validation of a Peer Support Specialist Checklist for Individuals With Opioid Use Disorder / STAMPS: South Carolina Buprenorphine Treatment Initiation, Adherence, and Retention Utilizing Mobile Health Units and Peer Support Specialists
Brief Title: STAMPS: South Carolina Buprenorphine Treatment Initiation, Adherence, and Retention Utilizing Mobile Health Units and Peer Support Specialists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2130836; R61DA059892-01 (NIH)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: peer support specialist; peer recovery coach; OUD; opioid use disorder; mobile health clinic; rural
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer Support Specialist Intervention (Experimental): Eligible participants will be linked to a peer support specialist. Peer support specialists are Certified Peer Support Specialists (CPSS) who have lived experience with opioid use disorder (OUD) and OUD recovery. Peer support specialists offer consistent personalized recovery support and generalized social support. Peer support specialists will maintain contact and provide support for the participant for 3 months post-baseline utilizing the newly validated checklist.
  Interventions: Behavioral: Peer Support Checklist

INTERVENTIONS:
Behavioral: Peer Support Checklist — Peer support specialists are Certified Peer Support Specialists (CPSS) who have lived experience with Opioid Use Disorder (OUD) and OUD recovery. Peer support specialists offer consistent personalized recovery support and generalized social support. Peer support specialists will maintain contact and provide support for the participant for six-months post-baseline. CPSS will utilize the newly developed checklist from earlier phases of the project to provide patient support.

SUMMARY:
The study is a 1-arm prospective interventional cohort quasi-experimental with retrospective control group. Enrolled participants will be compared to previously established mobile health patients, who did not work with a peer recovery coach, for buprenorphine treatment and adherence outcomes. 90 patients will be recruited from the mobile health units in rural counties in Upstate South Carolina. Visits consist of a baseline and 3 month follow up.

The study will focus to develop, deliver, and evaluate an innovative 1) Peer Support Specialist (PSS) intervention to increase Medications for Opioid Use Disorder (MOUD) initiation and retention rates in rural populations and underserved communities, and 2) dynamic modeling framework to prioritize at-risk communities for delivery of Mobile Health Clinics. the interventions will be developed in the R61 phase and implemented in a pilot study to determine the effectiveness on initiation and retention. With opioid overdose deaths continuing to rise in South Carolina (SC) and nationally, our sustainable framework has potential to prevent hundreds to thousands of opioid overdoses in SC and can be scaled up in other regions to save many more lives.

DETAILED DESCRIPTION:
Over 100,000 lives were lost due to drug overdose in the past year, of which 80% involved opioids.The majority of opioid-related deaths were due to fentanyl, an illicit opioid that has been labeled the single deadliest drug threat ever encountered in the United States.With opioid overdose deaths doubling in the past two years, there are no current signs that the epidemic is slowing down. Despite the effectiveness of medications for opioid use disorder (MOUD) at reducing opioid use, only 10% of those in need receive treatment. Furthermore, treatment retention is low (30-50%). Low treatment initiation and retention rates for Opioid Use Disorder (OUD) are especially concerning for rural and underserved communities, who rarely have access to clinicians prescribing MOUD and experience substantial barriers to care, including lack of insurance, social isolation, homelessness, transportation issues, and stigma. Given these populations are also at an elevated risk of overdose due to many of these same factors,interventions to increase MOUD initiation, retention, and overdose prevention in rural and underserved communities are urgently needed.

Our proposal aims to improve medication for opioid use disorder (MOUD) treatment rates and prevent overdose deaths in underserved communities using mobile health clinics (MHC). This will be achieved by developing, testing, delivering, and evaluating two key components: 1) a Peer Support Specialist (PSS) intervention to enhance MOUD initiation and retention, and 2) a modeling framework to identify high-risk communities for MHC delivery of opioid use disorder (OUD) interventions, based on the prevention of overdose deaths in those areas. Previous research has shown that such modeling tools can significantly enhance the efficiency of resource allocation across different health issues.

In the initial R61 phase, we will develop the PSS intervention and modeling framework.

The primary goal of aim 1 in the R61 phase is to assess the early fidelity, acceptability, and effectiveness of the PSS Service Delivery in boosting MOUD initiation and retention in rural and underserved populations. This intervention will draw from the successful assertive community engagement (ACE) model PSS interventions for substance use disorders and will be crafted based on qualitative interviews with PSS and OUD patients, as well as pilot data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Have diagnosis of OUD
* New patient of the mobile clinic

Exclusion Criteria:

* Currently prescribed MOUD
* Currently working with a PSS
* Current suicidal ideation, as verified through the Patient Health Questionnaire-9 (PHQ-9)
* Having a severe medical or psychiatric disability that would hinder participation in the study, as determined by nurse practitioner
* Unable to read/speak English
* Unable to read and comprehend the consent materials and other study materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Medication for Opioid Use Disorder (MOUD) Initiation | 3 months
  MOUD initiation is defined as receipt of first MOUD prescription within the 3-month study period
MOUD Retention | 3 months
  MOUD retention is defined as receipt of 75% of weekly MOUD prescriptions in first 3 months since MOUD initiation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Prisma Addiction Medicine Center - Mobile Health Clinic, Clinton, South Carolina
  - Prisma - Addiction Medicine Center Mobile Health Clinic, Seneca, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH RePORTER — https://reporter.nih.gov/project-details/10812747details